CLINICAL TRIAL: NCT00636922
Title: A Phase I Dose Finding Study of Everolimus (RAD001) in Elderly Patients With Acute Myeloid Leukemia (AML) Unfit for Intensive Induction Chemotherapy
Brief Title: Everolimus (RAD001) in Elderly Patients With Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C24112
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Elderly; Unfit; Everolimus; RAD001
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus with 5-azacitidine (Experimental): Everolimus increasing oral doses days 5-21 each cycle 5-azacitidine 75mg sub cutaneously 7 doses in 21 days
  Interventions: Drug: RAD001(Everolimus)

INTERVENTIONS:
Drug: RAD001(Everolimus) — In this study, 5-azacitidine will be administered sc for 7 doses over 9 days in a 28 day cycle. Everolimus will be administered orally with the first dose starting on day 5 (first Friday) of each cycle and continued until day 21 of each cycle. Patients will be treated with combined azacitidine + Everolimus for a minimum of 6 cycles and until at least 2 cycles after documentation of CR. Upon cessation of azacitidine, the patient will be permitted to take Everolimus maintenance therapy until progression at the investigator's discretion.
  Other Names: Everolimus

SUMMARY:
The main goal of this study is to assess the safety and tolerability of RAD001 in combination with low-dose cytarabine in acute myeloid leukemia patients unfit for intensive chemotherapy. The secondary goals are to investigate the likely causes of drug response or failure.

DETAILED DESCRIPTION:
A multicentre 2-stage Phase Ib/II trial of 5-Azacitidine combined with Everolimus for AML patients over the age of 60 or relapsed AML over the age of 18. The MTD and DLT of 5-Azacitidine (7 doses over 9 days) given monthly combined with Everolimus orally for 17 days (day 5-21) each month (1 cycle) for a minimum of 6 cycles and for at least 2 cycles beyond achievement of CR and for a maximum of 12 cycles. Everolimus maintenance therapy alone may be continued at investigator's discretion until either progressive disease or dose limiting toxicity. Groups of 3 patients will be entered at each dose level. Dose escalation/stopping rules to determine the maximum tolerated dose (MTD) are as follows:

Number in cohort experiencing DLT by day 42 Action 2/3 or 3/3 No further dose escalation. Previous level is defined as MTD 0/3 Dose escalate to next level 1/3 Expand cohort to 6 patients 1/6 or 2/6 Dose escalate to next level >2/6 No further dose escalation. Previous level is defined as MTD

Note that if dose escalation is still indicated at the highest dose level, then the MTD is at or above the last dose level. If the trial stops at the first dose, then the MTD is below the first dose level. In either of the above cases, the MTD is not determined from the trial.

Once the maximum dose level has been identified, a dose expansion phase will continue recruiting patients at the MTD until a total of 40 patients for the entire study is accrued.

ELIGIBILITY:
Untreated AML patients (defined by WHO 2008 criteria) over the age of 60 or relapsed/refractory AML over the age of 18 who have received up to 2 previous lines of intensive chemotherapy

* No prior failure to achieve at least a PR with Azacitidine or Everolimus
* Provision of written informed consent
* Secondary AML (including therapy-related) are included
* Life expectancy of greater than 3 months in relation to diseases other then AML/MDS
* ECOG performance status 0 - 3
* Electrolyte levels (potassium, calcium (albumin-adjusted), magnesium, phosphorous) within normal limits (WNL) or easily correctable with supplements
* Adequate hepatic function as defined by bilirubin ≤ 1.5 x the upper limit of normal (ULN) and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
* Adequate renal function, with serum creatinine ≤ 1.5 x ULN or GFR > 30 ml/minute
* Patients with no uncontrolled active infection
* Hydroxyurea ceased 48 hours prior to study therapy

Exclusion Criteria

* Any serious medical or psychiatric conditions which the investigator feels may interfere with the patient's ability to give informed consent or participate in the procedures or evaluations of the study
* History of major non-compliance to medication
* Evidence of CNS leukemia
* Uncontrolled viral infection with known HIV or Hepatitis type B or C
* Currently active gastrointestinal disease (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhoea, malabsorption syndrome, or small bowel resection), or other disease, that prevents the patient from absorbing or taking oral medication
* Any other concurrent severe and/or uncontrolled medical conditions (eg. acute or chronic liver disease, infection, pulmonary disease) that in the opinion of the investigator could potentiate unacceptable safety risks or jeopardize compliance with the protocol
* Males with a female partner of childbearing potential do not agree to use at least 2 effective contraceptive methods throughout the study and for 6 months following the date of last dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-02; Primary Completion 2013-07 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
safety & tolerability | over 24 cycles of treatment
  haematological toxicities (marrow status, neutrophil recovery), non-haematological grade 4 toxicity

SECONDARY OUTCOMES:
clinical Response | up to 3 years
  measure disease free survival up to 3 years
biomarkers of response | over length of treatment up to 24 cycles
  measure examples of biomarkers of disease response such as gene-specific methylation and phosphorylation status of mTOR targets
patient related outcomes | during treatment and in followup for up to 3 years
  Quality of life questionnaires and treatment related toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wei, MBBS PhD, Principal Investigator — Bayside Health
Locations (1):
- BaysideHealth, The Alfred Hospital, Melbourne, Victoria, Australia